CLINICAL TRIAL: NCT06213298
Title: Effect of Kava on Anxiety and Stress in Cancer Survivors
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Drug expiration testing
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HOT-2023-30373
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Kava; Anxiety; Stress; Cancer; Depression; Sleep
MeSH Terms: conditions — Anxiety Disorders; Neoplasms; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Kava (Experimental): 75mg of Kava taken three times daily for 14 days. Participants will then enter into a washout period of 14-28 days.
  Interventions: Drug: Kava
- Placebo (Placebo Comparator): The placebo will be taken three times daily for 14 days. Participants will then enter into a washout period of 14-28 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Kava — 75 mg kavalactones
  Arms: Kava
Dietary Supplement: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
This is a pilot, two-arm, randomized, blinded, placebo-controlled cross-over clinical trial to study the safety and effect of 14 days of kava on anxiety and physiologic stress in survivors of cancer and its treatment. Participants will be randomized to take either kava first or placebo first. Kava 75 mg or placebo will be taken three time daily (TID) for 14 days (Period 1), followed by a washout period of 14-28 days. Thereafter, the participant will take either placebo or kava TID for 14 days (Period 2), whichever he/she did not take in Period 1.

ELIGIBILITY:
Inclusion Criteria:

* Completed curative-intent treatment for breast, gynecologic, lung, or head/neck cancer within the last 24 months without clinical and/or radiographic evidence of recurrence at the time of the last follow up
* Score of ≥ 5 on the GAD-7 questionnaire, considered to be mild anxiety
* ECOG performance status 0-1
* Normal kidney and liver function within 28 days prior to the first dose of kava or placebo
* Willing to abstain from benzodiazepine and alcohol use during the kava or placebo intervention and for at least 14 days after completion
* Ability to provide written, informed consent

Exclusion Criteria:

* Regular use of benzodiazepines, defined as ≥ 2 times weekly, within 14 days prior to study registration
* Anti-cancer therapy within 28 days prior to registration, and/or during study participation, except for aromatase inhibitors
* Known liver disease such as cirrhosis (any Child-Pugh class), active infectious hepatitis, immune-mediated hepatitis, hemochromatosis, non-alcoholic steatohepatitis (NASH), or Wilson's disease
* Use of acetaminophen at doses more than 2000 mg daily for more than three days per week within 7 days prior to the first dose of kava or placebo intervention
* Chronic use of high-intensity statin therapy
* Significant uncontrolled conditions or situations, which in the judgment of the enrolling investigator, could affect safety and/or ability to adhere to study requirements
* Adjustments in anti-depressants and/or anxiolytic medications within 8 weeks prior to study registration
* Known allergy to kava
* Women who are pregnant, intend to become pregnant, or are nursing
* Regular use of alcohol, defined as ≥ 3 times per week, regardless of amount, within 14 days prior to study registration
* Parkinson's disease
* History of or current substance use disorder by self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in PROMIS anxiety measure score after 14 days of kava or placebo | 14 days
  PROMIS- 29 questionnaire will be administered to determine anxiety level. Scale 4-20. Higher score indicates higher anxiety.
Incidence of adverse events attributable to kava | 14 days
  Assessed using CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be shared amongst the study team via Box.